CLINICAL TRIAL: NCT02651532
Title: Confocal Endomicroscopy Utility for Diagnosing Mucosa Micro-inflammation in Patients With Irritable Bowel Syndrome
Brief Title: Confocal Endomicroscopy Utility (p-CLE) in Irritable Bowel Syndrome
Status: Completed | Type: Observational
Sponsor: Instituto Ecuatoriano de Enfermedades Digestivas (Other)
Responsible Party: Sponsor
Other Study IDs: ENE12016
Record Dates: First submitted 2016-01-07; First posted 2016-01-11 (Estimated); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Irritable Bowel Syndrome (IBS)
Keywords: Confocal Laser Endomicroscopy; inflammation; Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Histological biopsies of the colonic mucosal
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- IBS + Confocal Laser Endomicroscopy: Outpatients with irritable bowel syndrome according to Roma III classification: recurrent abdominal pain or discomfort, at least 3 days per month, in the last 3 months and symptoms begin at least 6 months before diagnosis, associated with 2 or more of: improvement with defecation, start associated with changes in the bowel frequency, start associated with changes in stool consistency. Absence of alarm symptoms: gastrointestinal bleeding, weight loss, anemia, night-time symptoms, fever, family history of colorectal cancer or celiac disease, elevated erythrocyte sedimentation rate, positive fecal occult blood test.
  Interventions: Device: Confocal Laser Endomicroscopy
- Control + Confocal Laser Endomicroscopy: Outpatients without IBS symptoms, undergoing colonoscopy for colorectal cancer screening
  Interventions: Device: Confocal Laser Endomicroscopy

INTERVENTIONS:
Device: Confocal Laser Endomicroscopy — During colonoscopic withdrawal, the colonic mucosa will be observed with white light and be evaluated on the different segments of the colon with the confocal laser endomicroscopy technology in order to search for microscopic inflammation signs (altered crypt architecture, fluorescein leaks and dilated and prominent branching vessels)

SUMMARY:
Irritable bowel syndrome (IBS) is one of the most common gastrointestinal disorders. It has prevalence in general population of 5-20% and is more common in women and young adults.

Despite being one of the most frequent reasons for consultation many patients are undiagnosed. There are no reliable biomarkers. The diagnosis is clinical, based on the Rome III criteria. IBS is characterized by chronic or recurrent abdominal pain associated with changes in bowel frequency and consistency, when other etiologies are excluded. The combination of the Rome III criteria with the absence of alarm symptoms have a sensitivity of 65%, specificity of 100%, 100% positive predictive value and negative predictive value of 76%.

Current tests commonly fail to obtain an objective diagnosis, and effective therapies are lacking. There are no specific endoscopic findings that can discriminate IBS patients from healthy patients. Most colonoscopies are performed to rule out other etiologies and in more than 50% of the cases are normal.

DETAILED DESCRIPTION:
The pathophysiology is complex, multifactorial and not completely known. Impaired intestinal barrier function and mucosal inflammation in the small and large intestine have been reported. Evidence of inflammation and neuronal degeneration in the myenteric plexus has been found in full-thickness intestinal biopsy samples from IBS patients.

It has been found that IBS patients had a significantly higher density of intestinal epithelial gaps. The elevated epithelial gaps in the intestine of IBS patients, a surrogate marker for increased epithelial cell extrusion, may be a cause of altered intestinal permeability observed and may lead to mucosal inflammation.

Confocal laser endomicroscopy (CLE) is a new endoscopic imaging tool enabling visualization of changes in the gut mucosa. The use of intravenous fluorescein enables high-resolution real-time imaging in vivo at a micron scale, allowing visualization of cellular details during ongoing endoscopy. This technology can be used to identify and quantify epithelial gaps and other signs of inflammation.

The purpose of this study is to evaluate the presence of microscopic inflammation previously demonstrated in patients with IBS, using pCLE. The determination of the exact areas of inflammation allows a direct biopsy in a more accurate way. This type of systematic may allow in the future to classify these patients not only symptomatically (constipation, diarrhea or mixed predominant IBS) but also according to their degree of inflammation. There is no Gold Standard test in these patients to assess response to treatment. The possibility of using pCLE to identify the areas of microscopic inflammation allows that the degree of inflammation can be used as a monitoring parameter. Probably the CLE can be used to assess response to treatment and different types of treatments, determining differences between subtypes of patients with IBS, evaluate remission, recurrence and prognosis. Also it may clarify a potential mechanism of the pathogenesis and be endoscopic criteria for the diagnosis of the disease.

The present study is the first to evaluate the colon microscopic inflammation using pCLE in IBS patients.

Study design: This is an observational and analytical cross-section, population - based survey study, with prospective case collection, non-randomized and simple blind, performed in a Tertiary Academic Center.

Setting: Ecuadorian Institute of Digestive Diseases (IECED), OmniHospital Academic Tertiary Center. We will include patients from October 2015 to March 2016. Patients will be recruited from the gastroenterology unit (IECED). The study protocol and consent form has been approved by the Institutional Review Board (IRB) and will be conducted according to the declaration of Helsinki. Patients will sign an informed consent and answer a questionnaire that includes constitutional data (sex, age, comorbid medical condition, medication). Patients in IBS group will be classified according to the symptoms as diarrhea predominant (IBS-D), constipation predominant (IBS-C) or mixed type (IBS-M). Endoscopic findings will be recorded in a database.

Endoscopic technique: All colonoscopies will be performed after the patient had undergone standard bowel preparation using either polyethylene glycol electrolyte lavage solution. Initially a routine white light colonoscopy will be performed in IBS and healthy control patients, using a Pentax scope (Pentax EC-387CILK, Tokyo, Japan) with great care not to damage the epithelium. The Boston Bowel Preparation Scale and inflammation changes will be recorded.

During withdrawal, all parts of the colon will be evaluated (cecum, right-side colon, transverse, left-side colon, sigmoid and rectum) using pCLE randomly in one point of each segment, if there are no signs of iatrogenic mucosal damage. Careful washing of the mucosa with water in order to prevent the inclusion of image artefacts from residual stool fragments. Before initiating CLE evaluation, intravenous injection of 5 ml 10% fluorescein will be done. Fluorescein stains vessels and gives good tissue structure, but the nuclei are not stained and appear as dark spots. Optimal contrast is obtained within the first 10min after injection, but good quality images can be acquired for a further 30-60 min.

Currently Confocal Laser Endomicroscopy (CLE) is performed using a CLE probe (pCLE). The confocal microscope used in pCLE captures microscopic images of untreated in vivo tissue. The microscope uses focused laser light of a defined wavelength and passes it through a confocal aperture. Images are then reconstructed in two dimensions. For pCLE (Cellvizio by Mauna Kea Technologies, Paris, France), both the laser scanning unit and light source are outside the body. The laser beam is transported via flexible confocal miniprobes and a distal lens sequentially scans it through a bundle of more than 10000 optical fibers. Confocal miniprobes are flexible, with diameters ranging from 0.9 mm to 2.5 mm.

In the study a pCLE ColoFlex probe will be used (Cellvizio; Mauna Kea Technology, Paris, France). The probe goes through the accessory channel of a conventional endoscope. The image rate is 0.08 s/frame at 1024×1024 pixels with a imaging depth of 20 μm. The confocal images will be first analyzed during the endoscopy. Then, the images will be digitally stored and reviewed after the procedure in order to zoom in on details for a higher magnification (approximately 10000 fold), with special designed software package (Cellvizio Viewer), allowing image correction and stabilization.

Immediately after pCLE evaluation, and before proceeding to the next colon segment, targeted biopsies will be taken from the mucosal area evaluated. Bleeding can impair image quality, therefore probe will be placed gently in contact with the tissue in order to avoid trauma and pCLE imaging will be completed in a region before mucosa biopsy. The endoscopist performing the pCLE will be blinded to the status of the patient and the images will be later analyzed in detail blindly by two different persons with more than two years' experience in endomicroscopy.

There are not studies that validate a classification of colon inflammation using CLE in IBS patients. Inflammation of the colon mucosa in ulcerative colitis (UC) has been described previously using CLE. Kiesslich et al. reported on a 3-grade classification of inflammation activity by CLE, combining crypt architecture, cellular infiltrations, and vessel architecture. Nevertheless the assessment of cellular infiltration has been questioned because of the difficulty in differentiating cell types by CLE. Chang-Qing Li, et al. used three CLE parameters to evaluate inflammation in UC patients: a 4-grade crypt-architecture classification, fluorescein leakage, and microvascular alterations. On the other hand, the Miami classification for pCLE defines colitis using: crypt fusion and distortion, bright epithelium, dilated and prominent branching vessels.In the present study the parameters used for CLE inflammation will be: 1.Epithelial gaps followed by leaks with secretion of fluorescein into the lumen. In CLE images of normal colonic mucosa, the lumen of the crypt is free of fluorescein and appears as a dark center in the crypt; however, in inflamed mucosa, fluorescein leaks into the crypt lumen; therefore, the lumen is brighter than the surrounding epithelium. 2.4-grade crypt-architecture classification: Types A and B will be considered as normal and chronic inflammation, respectively, and types C and D indicate acute inflammation. Type A: Regular arrangement and size of crypts. Type B: Irregular arrangement of crypts, enlarged spaces between crypts. Type C: Dilation of crypt openings, more irregular arrangement of crypts, and enlarged spaces between crypts as compared to type B. Type D: Crypt destruction and / or crypt abscess. 3.Dilated and prominent branching vessels

Interobserver and Intraobserver Agreement: A data set containing CLE photographs and videos of the all of the colon segments will be presented to three blinded endoscopists, who will confirm or not the findings. Inter- and intra-observer reproducibility will be measured based on comparison of still images and videos between the three investigators. To evaluate the intra-observer agreement each investigator will assess the images two times and the answers will be compared. To evaluate the inter-observer agreement all answers between the three investigators will be compared. In general, the learning curve of CLE is short and inter or intra-observer agreement is good.

Statistical analysis: Baseline characteristics will be compared between case and control group using Chi-square o Fisher Test for categorical variable, and for continuing variables, we will use the Mann-Whitney Test. Diagnosis efficacy will be measured thought sensitive, specificity and accuracy. All the statistical analysis will be performed using SPSS software suite v.22.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old patients
* Who agree to participate in the study
* Ability to provide written informed consent
* Patients with irritable bowel syndrome according to Roma III classification.

Exclusion Criteria:

* Patients, who were receiving nonsteroidal anti-inflammatory drugs, corticosteroids or antibiotics in the last 4 weeks.
* Patients with heart disease, kidney, liver or severe metabolic disorder, who cannot tolerate sedation
* Inflammatory bowel disease
* Bacterial overgrowth
* Gastrointestinal bleeding
* Prior history of any king of colitis (actinic, infectious, ischemic, microscopic colitis)
* Suspected colonic obstruction or history of previous obstruction
* Prior history of colectomy surgery
* Patients with an ileostomy or a colostomy
* Patients with difficulty understanding instructions of bowel preparation
* Known allergy to fluorescein or shellfish
* Pregnancy and lactation
* Bowel preparation will be evaluated using the Boston Bowel Preparation Scale. (9) Patients with < 2 points in at least one of the three segments of the colon (rectum plus left-side colon, transverse colon plus left and right flexure, right-side colon) will be excluded from statistical analysis as well as those who after the beginning of the colonoscopy, had to be aborted because of an inability to reach the cecum by unfavorable anatomy or impassable tumors / stenosis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients with irritable bowel syndrome according to Roma III classification: recurrent abdominal pain or discomfort, at least 3 days per month, in the last 3 months and symptoms begin at least 6 months before diagnosis, associated with 2 or more of: 1) Improvement with defecation, 2) Start associated with changes in the bowel frequency, 3) Start associated with changes in stool consistency. In the absence of alarm symptoms. It will be measured in all patients serology for celiac disease, serum thyroid-stimulating hormone (TSH) and parasitological test. It will be done, in high suspicion patients, stool culture, breath test for lactose intolerance and breath test for bacterial overgrowth.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2016-01; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Confocal Laser Endomicroscopy (CLE) utility for diagnosing microscopic inflammation of the mucosa in patients with irritable bowel syndrome (IBS) | four month
  Number of patients with IBS and microscopic inflammation determinate by CLE

SECONDARY OUTCOMES:
Relationship between microscopic inflammation and sex, age and the subtypes of IBS. | four month
  Number of patients with microscopic inflammation according to sex, age and the subtypes of IBS.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Robles-Medranda, MD, Principal Investigator — Ecuadorian Institute of Digestive Diseases
Locations (1):
- Ecuadorian Institute of Digestive Diseases, Guayaquil, Guayas, Ecuador

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Longstreth GF, Thompson WG, Chey WD, Houghton LA, Mearin F, Spiller RC. Functional bowel disorders. Gastroenterology. 2006 Apr;130(5):1480-91. doi: 10.1053/j.gastro.2005.11.061. PMID 16678561
- [Result] Drossman DA. The functional gastrointestinal disorders and the Rome III process. Gastroenterology. 2006 Apr;130(5):1377-90. doi: 10.1053/j.gastro.2006.03.008. No abstract available. PMID 16678553
- [Result] Mayer EA. Clinical practice. Irritable bowel syndrome. N Engl J Med. 2008 Apr 17;358(16):1692-9. doi: 10.1056/NEJMcp0801447. PMID 18420501
- [Result] Drossman DA, Camilleri M, Mayer EA, Whitehead WE. AGA technical review on irritable bowel syndrome. Gastroenterology. 2002 Dec;123(6):2108-31. doi: 10.1053/gast.2002.37095. No abstract available. PMID 12454866
- [Result] Tornblom H, Lindberg G, Nyberg B, Veress B. Full-thickness biopsy of the jejunum reveals inflammation and enteric neuropathy in irritable bowel syndrome. Gastroenterology. 2002 Dec;123(6):1972-9. doi: 10.1053/gast.2002.37059. PMID 12454854
- [Result] Kiesslich R, Goetz M, Angus EM, Hu Q, Guan Y, Potten C, Allen T, Neurath MF, Shroyer NF, Montrose MH, Watson AJ. Identification of epithelial gaps in human small and large intestine by confocal endomicroscopy. Gastroenterology. 2007 Dec;133(6):1769-78. doi: 10.1053/j.gastro.2007.09.011. Epub 2007 Sep 16. PMID 18054549
- [Result] Turcotte JF, Kao D, Mah SJ, Claggett B, Saltzman JR, Fedorak RN, Liu JJ. Breaks in the wall: increased gaps in the intestinal epithelium of irritable bowel syndrome patients identified by confocal laser endomicroscopy (with videos). Gastrointest Endosc. 2013 Apr;77(4):624-30. doi: 10.1016/j.gie.2012.11.006. Epub 2013 Jan 26. PMID 23357497
- [Result] Fritscher-Ravens A, Schuppan D, Ellrichmann M, Schoch S, Rocken C, Brasch J, Bethge J, Bottner M, Klose J, Milla PJ. Confocal endomicroscopy shows food-associated changes in the intestinal mucosa of patients with irritable bowel syndrome. Gastroenterology. 2014 Nov;147(5):1012-20.e4. doi: 10.1053/j.gastro.2014.07.046. Epub 2014 Jul 30. PMID 25083606
- [Result] Lai EJ, Calderwood AH, Doros G, Fix OK, Jacobson BC. The Boston bowel preparation scale: a valid and reliable instrument for colonoscopy-oriented research. Gastrointest Endosc. 2009 Mar;69(3 Pt 2):620-5. doi: 10.1016/j.gie.2008.05.057. Epub 2009 Jan 10. PMID 19136102
- [Result] Kuiper T, Kiesslich R, Ponsioen C, Fockens P, Dekker E. The learning curve, accuracy, and interobserver agreement of endoscope-based confocal laser endomicroscopy for the differentiation of colorectal lesions. Gastrointest Endosc. 2012 Jun;75(6):1211-7. doi: 10.1016/j.gie.2012.01.040. Epub 2012 Mar 28. PMID 22459661
- [Result] Wallace M, Lauwers GY, Chen Y, Dekker E, Fockens P, Sharma P, Meining A. Miami classification for probe-based confocal laser endomicroscopy. Endoscopy. 2011 Oct;43(10):882-91. doi: 10.1055/s-0030-1256632. Epub 2011 Aug 4. PMID 21818734
- [Result] Becker V, von Delius S, Bajbouj M, Karagianni A, Schmid RM, Meining A. Intravenous application of fluorescein for confocal laser scanning microscopy: evaluation of contrast dynamics and image quality with increasing injection-to-imaging time. Gastrointest Endosc. 2008 Aug;68(2):319-23. doi: 10.1016/j.gie.2008.01.033. Epub 2008 Apr 24. PMID 18436217
- [Result] Kiesslich R, Goetz M, Lammersdorf K, Schneider C, Burg J, Stolte M, Vieth M, Nafe B, Galle PR, Neurath MF. Chromoscopy-guided endomicroscopy increases the diagnostic yield of intraepithelial neoplasia in ulcerative colitis. Gastroenterology. 2007 Mar;132(3):874-82. doi: 10.1053/j.gastro.2007.01.048. Epub 2007 Jan 31. PMID 17383417
- [Result] Li CQ, Xie XJ, Yu T, Gu XM, Zuo XL, Zhou CJ, Huang WQ, Chen H, Li YQ. Classification of inflammation activity in ulcerative colitis by confocal laser endomicroscopy. Am J Gastroenterol. 2010 Jun;105(6):1391-6. doi: 10.1038/ajg.2009.664. Epub 2009 Nov 24. PMID 19935787